CLINICAL TRIAL: NCT04955600
Title: Introducing Technology in the Home of Elderly Patients With Multimorbidity, a Hybrid Effectiveness Implementation Study
Brief Title: Digital Technology in the Home of Elderly Patients With Multimorbidity
Status: Completed | Type: Observational
Sponsor: Sormland County Council, Sweden (Other)
Collaborators: Swedish Association of Local Authorities and Regions (Other)
Responsible Party: Principal Investigator, Maria Liljeroos, Principal Investigator, Sormland County Council, Sweden
Other Study IDs: Maria Liljeroos
Record Dates: First submitted 2021-06-16; First posted 2021-07-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Multimorbidity
Keywords: telemonitoring; distance monitoring; feasibility; implementation; elderly

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients with multimorbidity, relatives, health care personal: The care team consists of four nurses, two of whom are employed by the region and two by the municipality, 20 municipally employed assistant nurses and one physician. Other professions associated with the team are psychologist, dietitian, pharmacist, counsellor, physiotherapist, occupational therapist, and family consultants. All participants in the team will be invited to participate in the study. The technology will be place in 20-25 patients' home and patients and family members will be invited to participate in the study. Self-care education will be given to the patients and family members according to the middle-range theory of self-care of chronic illness.
  Interventions: Other: Implementation Study

INTERVENTIONS:
Other: Implementation Study — Implementation of digital technology in two different care settings from both patients, informal caregivers, and healthcare professional's perspective.

SUMMARY:
In this study, the objective is to evaluate available technology designed to support self-care at home of elderly patients with multimorbidity. Of people who are 85 years or older, about 60% have two or more chronic diseases. The symptom burden is extensive, and periods of deterioration often lead to hospitalizations and early readmissions to hospital. A contributing factor for the high consumption of care is that many patients find it difficult to identify signs of deterioration and in time take appropriate action. Technology placed in patients' home are becoming common and have shown to increase quality of life and reduce the need for in-hospital care but few tools are used in regular care.

The investigators want to see which effect technologies placed at home has on; healthcare consumption, self-care, depression, well-being and activity level. Further, the implementation process from both patients, relatives and healthcare personals perspective will be studied using a hybrid design, which makes it possible to study both barriers and facilitators of the implementation and efficacy of the technology.

In phase one participants will be recruited from a care team where an established collaboration between region and municipality has been developed. In phase two, inclusion takes place in an entire municipality without a previously established collaboration. The goal is to increase patients and family members wellbeing, health and functional ability while maintaining or reducing healthcare costs.

DETAILED DESCRIPTION:
PURPOSE AND AIMS In this study, the objective is to evaluate available digital technology with remote symptom monitoring designed to support self-care at home of elderly patients with multimorbidity. There are a lot of technology with the possibility to remotely monitor signs and symptoms placed in patients' home available. This technology have been shown to increase quality of life, experiences of security and reduce the need for in-hospital care, but few tools are implemented in routine care of elderly with multimorbidity and extensive needs of coordinated health and community care. Limited collaboration and lack of joint care goals between the different care providers are known barriers of implementation of digital technology with remote symptom monitoring.

The overall aims of the project are:

1. To describe the implementation process of digital technology in two different care settings from both patients, family members, and healthcare professional's perspective.
2. To evaluate the feasibility of digital technology for remote symptom monitoring and digital consultations with the caregiver in the home of elderly patients with multimorbidity.
3. To examine the effectiveness of the technology.

Specific research questions the study is set to answer:

1. What effects does the use of digital technology for remote symptom monitoring have on elderly patients with multimorbidity's healthcare consumption, self-care management, depression, experience of control over the disease, well-being and activity level?
2. How do patients and informal caregivers perceive that the use of digital technology at home affects the ability to manage the patient's health situation?
3. How do physicians, nurses and assistant nurses experience the use of remote monitoring in their daily work?
4. Which are the barriers to and facilitators for implementation of digital technology?
5. Does digital technology reduce the risk of hospitalisation and healthcare costs in elderly patients with multimorbidity?

The study has a hybrid design, which means a double focus: both the implementation process and the clinical outcomes are studied simultaneously through a mixed data collection with both quantitative and qualitative parts. The implementation process will be based on The Quality Implementation Framework.

Phase 1; During winter 2021-22 the implementation process of digital technology with remote symptom monitoring with adaptation and preparation in the care team will begin. The team needs to develop a structure for handling the incoming patient data and develop action plans on how to act in case of symptoms and signs of deterioration.

The technology, OPTILOGG PLUS, will be place in patients' home.It consists of a tablet with personalized sensors, such as weighing scale, blood pressure, oxygenation and activity meters based on the patient's individual needs. The technology also includes a platform for digital consultation.

The patient performs measurements at home every morning and sends data to the receiving station installed in the care teams' premises where the staff access the patient's data via secure login.The main purpose of the technology is to enhance the patients' self-care behaviour, and coach them to contact the healthcare provider if and when self-care is not enough to prevent deterioration. Also the caregiver can initiate a virtual home visit or a physical home visit if they observe signs of deterioration not recognised by the patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in the care team and their family members who will have digital technology placed in their home will be asked to participate.
* All healthcare personal in the care team will be asked to participate

Exclusion Criteria:

* 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to include all patients, family members and healthcare personal who is involved in the process of implementation of digital technology.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of digital technology | December 2021-December 2022
  Healthcare consumption will be performed via regions healthcare database.
Implementation process | April 2021-December 2021
  Healthcare professionals will be asked about potential barriers and facilitators for implementation of the technology, problems associated with the implementation, potential modifications that could be made to maximize implementation, potential implementation strategies, skills or training necessary for healthcare professionals to work with the technology.

SECONDARY OUTCOMES:
Experience of digital technology | December 2021-December 2022
  Experience of the technology will be measured by a self-designed survey. Care and nursing staff from both the region and the municipality will is asked to answer a self-constructed questionnaire regarding experiences of the implementation of digital technology,
Anxiety and depression | December 2021-December 2022
  In-depth surveys for patients; Hospital Anxiety and Depression Scale
Perceived control | December 2021-December 2022
  Control Attitude Scale
Well-being | December 2021-December 2022
  WHO Welfare Index
Physical activity | December 2021-December 2022
  Frändin Grimby's activity scale

CONTACTS AND LOCATIONS:
Locations (1):
- Care team in Region of Sörmland, Eskilstuna, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liljeroos M, Arkkukangas M, Stromberg A. The long-term effect of an m-health tool on self-care in patients with heart failure: a pre-post interventional study with a mixed-method analysis. Eur J Cardiovasc Nurs. 2024 Jul 19;23(5):470-477. doi: 10.1093/eurjcn/zvad107. PMID 38165027